CLINICAL TRIAL: NCT00257504
Title: Registration of Central Blood Volume in Hypotensive Dialysis Patients - a Comparison of Thoracic Impedance and Central Venous Saturation Monitoring
Brief Title: Central Blood Volume in Hypotensive Dialysis Patients
Status: Completed | Type: Observational
Sponsor: Danish State Hospital (Other)
Other Study IDs: CBV estimation
Record Dates: First submitted 2005-11-21; First posted 2005-11-23 (Estimated); Last update posted 2006-09-12 (Estimated); Status verified 2006-09

CONDITIONS: Intradialytic Hypotension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
The purpose of the study is to test whether hypotensive episodes during dialysis - caused by withdrawal of fluid drom the circulation - can be predicted by means of two harmless monitoring techniques.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis patients with central vascular access

Exclusion Criteria:

* Patients below 18 years of age
* Patients unable to give informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-11; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: Søren D Ladefoged, MD, Study Director — Danish State Hospital
Locations (1):
- Danish State Hospital, Copenhagen, Denmark